CLINICAL TRIAL: NCT00540111
Title: Effect of Soluble Fiber on Hypertriglyceridemia and Immune Profile in HIV-positive Individuals on Highly Active Antiretroviral Therapy
Brief Title: Effect of Soluble Fiber on Hypertriglyceridemia and Immune Profile in HIV-positive Individuals.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Botucatu Medical School - UNESP, Juliana Geraix
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-01
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Hypertriglyceridemia; HIV Infections
Keywords: Soluble fiber; HIV/aids; Hypertriglyceridemia; Cytokines; Alternative Medicine; Complementary Medicine
MeSH Terms: conditions — Hypertriglyceridemia; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — lactitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Study of intervention, prospective,uncontrolled Group Number: 1
  Group Type:Other - the subjects of group were compared the initial moment (M0 - moment without soluble fiber supplementation)with the others two moments: M1 (one month after soluble fiber supplementation) and M2 (four months after soluble fiber supplementation).
  Group Description - HIV-positive individuals with hypertriglyceridemia (serum levels ≥ 200 to ≤ 500 mg/dL),who had been on the same HAART regimen for at least 6 months, had no change in therapy during the study.
  Intervention:Received 20g/day of soluble fiber® (partially hydrolyzed guar gum) for 4 months at pre-established times.
  Interventions: Dietary Supplement: soluble fiber® (partially hydrolyzed guar gum)

INTERVENTIONS:
Dietary Supplement: soluble fiber® (partially hydrolyzed guar gum) — HIV-positive individuals with hypertriglyceridemia and who had been on the same HAART regimen for at least 6 months, had no change in therapy during the study,received 20g/day of soluble fiber for 4 months at pre-established times.
  Other Names: Benefiber® (Novartis)

SUMMARY:
The purpose of this study was to assess the effect of soluble fiber® (partially hydrolyzed guar gum) supplementation on hypertriglyceridemia and immune profile in HIV-positive individuals on HAART.

DETAILED DESCRIPTION:
Since 1996, the advent of highly active antiretroviral therapy (HAART) has caused a profound impact on the natural history of HIV-infection by promoting important and sustainable viral replication suppression and increasing survival and quality of life among seropositive patients. Nonetheless, antiretroviral therapy has been observed to be accompanied by metabolic alterations such as dyslipidemia, especially hypertriglyceridemia, insulin resistance, hyperglycemia and lipodystrophy (body fat redistribution). Epidemiological studies have demonstrated a correlation between high triglyceride (TG) levels and higher incidence of coronary artery disease (CAD). Some investigators suggest dietary intervention as part of hyperlipidemia treatment, including an increase in soluble fiber intake (10-25g/day). Whereas some studies have demonstrated that both cholesterol and serum triglyceride levels decrease with the use of food fiber, others have shown just a serum triglyceride increase, and others failed to observe any alteration in lipid metabolism. The purpose of this study was to assess the effect of soluble fiber® (partially hydrolyzed guar gum) supplementation on hypertriglyceridemia and immune profile in HIV-positive individuals on HAART. Nineteen HIV-positive individuals with hypertriglyceridemia (serum levels ≥ 200 to ≤ 500 mg/dL) were studied. Of these individuals, 63.16% were males (mean age of 38.52±9.29 years) who had been on the same HAART regimen for at least 6 months, had no change in therapy during the study and received 20g/day of soluble fiber for 4 months at pre-established times. Clinical-nutritional, biochemical (total proteins, albumin, globulin, total cholesterol, LDL-c, HDL-c, TG, TG/HDL-c and LDL-c/HDL-c), hemoximetric (hemoglobin, hematocrit and total lymphocytes), and immunologic (lymphocytes T CD4+, T CD8+; T CD4+/CD8+ ratio, viral load, TNFα- and IL-6) parameters were assessed in all patients at three time points (M0-pretreatment, M1-30 days and M2-4 months after intervention). Significance level was set 5% for all data statistically analyzed. Serum TG and TG/HDL-c ratio reduction was observed at all time points, but statistical significance was found just at M0 and M2. The remaining biochemical, hemoximetric and immunologic parameters (lymphocytes T CD4+, T CD8+; T CD4+/CD8+ ratio, and viral load) showed no significant difference at all times. Regarding serum cytokines, TNFα- and IL-6 significantly decreased between M0 and M2, and only IL-6 reduced between M1 and M2. The data collected show that dietary and anthropometric parameters remained unchanged excluding potential confounding factors related with the effect of fiber supplementation on serum TG, TNFα- and IL-6. Thus, soluble fiber® (partially hydrolyzed guar gum) contributed to an important reduction in hypertriglyceridemia and in the serum levels of the proinflammatory cytokines TNFα- and IL-6 in HIV-seropositive individuals on HAART. In addition, soluble fiber® (partially hydrolyzed guar gum) might have minimized the process of atherosclerosis in these individuals, given that elevated serum levels of TG, TNFα- and IL-6 have been associated with the development of these lesions.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of HIV
* Hypertriglyceridemia
* Use of highly active antiretroviral therapy

Exclusion Criteria:

* Use of hypolipemic drugs
* Use of highly active antiretroviral therapy under six months
* Pregnant
* Insulin independent diabetes
* Thyroid disease
* Others infectious
* Alcoholic
* Under 18 years old

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2005-03; Primary Completion 2007-07 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Serum TG and TG/HDL-c ratio reduction was observed at all time points, but statistical significance was found just at M0 and M2. Regarding serum cytokines, TNFα- and IL-6 significantly decreased between M0 and M2, and only IL-6 reduced between M1 and M2. | four months

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Geraix, Nutricionist, Principal Investigator — Botucatu Medical School - UNESP; Paulo CM Pereira, PhD, Study Chair — Botucatu Medical School - UNESP